CLINICAL TRIAL: NCT04576806
Title: Physiological Effects of 38°C vs. 22°C Fluid Therapy in Critically Ill Patients: A Randomized Controlled ICU Study
Brief Title: Physiological Effects of 38°C vs. 22°C Fluid Therapy in Critically Ill Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Other research priorities during Covid-19 pandemic.
Sponsor: Karolinska Institutet (Other)
Collaborators: Danderyd Hospital (Other); Stockholm South General Hospital (Other)
Responsible Party: Principal Investigator, Christer Svensen, Clinical Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EPN 2019-05492
Record Dates: First submitted 2020-02-23; First posted 2020-10-06 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Critical Illness; Sepsis; Fluid Overload; Hemodynamic Instability
Keywords: Fluid therapy; Bolus
MeSH Terms: conditions — Critical Illness; Sepsis; Edema | interventions — Body Temperature

STUDY DESIGN:
Intervention Model Description: RCT, unblinded
Who Masked: Outcomes Assessor
Masking Description: Investigators will be blinded during analysis but unblinded during study performance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Body temperature fluid bolus of crystalloid (Active Comparator): Fluid bolus at 38 degrees celsius of 500ml crystalloid over 15 minutes
  Interventions: Other: Body temperature; Drug: Fluid bolus
- Room temperature fluid bolus of crystalloid (Experimental): Fluid bolus at 22 degrees celsius of 500ml crystalloid over 15 minutes
  Interventions: Drug: Fluid bolus; Other: Room temperature

INTERVENTIONS:
Other: Body temperature — Warming of administered fluid bolus
  Arms: Body temperature fluid bolus of crystalloid
Drug: Fluid bolus — Administration of fluid bolus of crystalloid of 500ml over 15 minutes
Other: Room temperature — Cooling of administered fluid bolus
  Arms: Room temperature fluid bolus of crystalloid

SUMMARY:
A randomized controlled clinical trial. 24 adult ICU patients will be recruited upon decision to administer fluid bolus of 500ml of crystalloid. The fluid will then be randomized to be infused at controlled room temperature or warmed to body temperature. Hemodynamic measurements will be made for 2 hours following the bolus, and laboratory values will be noted. The hypothesis is that part of the hemodynamic response will differed in response to cooling, and be larger in the cold group.

DETAILED DESCRIPTION:
A randomized controlled clinical trial of the influence of fluid temperature on hemodynamic effects of fluids. 24 adult ICU patients meeting objective criteria of circulatory impairment (hypotension, tachycardia, lactatemia etc) will be recruited upon decision to administer fluid bolus of 500ml of crystalloid. The fluid will then be randomized to be infused at controlled room temperature of 22 degrees or warmed to body temperature at 38 degrees. All patients will be monitored with either calibrated or uncalibrated pulse contour analysis. Hemodynamic measurements (Heart rate (HR), Systolic blood pressure (SBP), Diastolic blood pressure (DBP), Mean arterial pressure (MAP), Cardiac output (CO), Cardiac index (CI), Stroke volume (SV), Stroke volume variation (SVV), Extravascular lung water (EVLW) etc) will be registered for 2 hours following the bolus, and laboratory values such as lactate, creatinine will be noted, as well as fluid balances. Confounders such as levels of vasopressors, sedation, switches in positioning och or ventilation will be registered. The hypothesis is that part of the hemodynamic response will differed in response to cooling, and be larger in the cold group.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the ICU
* Age 18 years or older
* Clinical decision to administer a fluid bolus of at least 500 ml of crystalloid over 15 minutes.
* Monitoring with either an arterial line in an extremity that can be used for pulse contour analysis (Vigileo, FloTrac or equivalent system) or a central venous catheter and a femoral arterial line that can be used for pulse contour analysis calibrated by thermodilution (EV1000, PiCCO or equivalent system)
* At least one of the following criteria for fluid administration must be met:
* MAP < 65 mmHg
* HR >100
* Urine output < 0,5ml/kg/h
* Lactate levels of > 3 mmol/l
* CI < 2.5L/min/m2
* SVV or PPV > 12% if mechanically ventilated with tidal volumes > 7 ml/kg
* ScvO2 or SvO2 < 65%

Exclusion Criteria:

* Active bleeding requiring transfusion
* Haemoglobin level <70 g/L
* Arrhythmia disturbing monitoring of cardiac output
* Patients in whom death is considered imminent (within 24 hours)
* CRRT
* Known pregnancy
* Active temperature control, either active warming or cooling
* Medical issue of pathological thermoregulation, such as malignant hyperthermia, thyroid storm, NMDA overdose, serotonin syndrome, malignant neuroleptic syndrome, or delirium.
* Planned exit from the ICU during the 2-hour monitoring period (planned surgical procedure, radiology, change of department etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-30 (Estimated); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
MAP | 15 minutes
  Mean arterial pressure

SECONDARY OUTCOMES:
MAP | 1 hour
  Systolic blood pressure
MAP | 2 hours
  Systolic blood pressure
SBP | 15 minutes
  Systolic blood pressure
SBP | 1 hour
  Systolic blood pressure
SBP | 2 hours
  Systolic blood pressure
DBP | 15 minutes
  Diastolic blood pressure
DBP | 1 hour
  Diastolic blood pressure
DBP | 2 hours
  Diastolic blood pressure
HR | 15 minutes
  Heart rate
HR | 1 hour
  Heart rate
HR | 2 hours
  Heart rate
CO | 15 minutes
  Cardiac output
CO | 1 hour
  Cardiac output
CO | 2 hours
  Cardiac output
CI | 15 minutes
  Cardiac index
CI | 1 hour
  Cardiac index
CI | 2 hours
  Cardiac index
SV | 15 minutes
  Stroke volume
SV | 1 hour
  Stroke volume
SV | 2 hours
  Stroke volume
SVV | 15 minutes
  Stroke volume variation
SVV | 1 hour
  Stroke volume variation
SVV | 2 hours
  Stroke volume variation
EVLW | 15 minutes
  Extra vascular lung water
EVLW | 1 hour
  Extra vascular lung water
EVLW | 2 hours
  Extra vascular lung water
Type ofh eart rhythm | 15 minutes
  Heart rhythm
Type of heart rhythm | 1 hour
  Heart rhythm
Type of heart rhythm | 2 hours
  Heart rhythm
Levels of administered vasopressors | 15 minutes
  Amount of pressors
Levels of administered vasopressors | 1 hours
  Amount of pressors
Levels of administered vasopressors | 2 hours
  Amount of pressors
Levels of administered sedating medications | 15 minutes
  Amount of sedation
Levels of administered sedating medications | 1 hours
  Amount of sedation
Levels of administered sedating medications | 2 hours
  Amount of sedation
Lactate | 15 minutes
  Lactate
Levels of lactate | 1 hour
  Lactate
Levels of lactate | 2 hours
  Lactate
Hourly urine output | 1 hour
  Urine output
Hourly urine output | 2 hours
  Urine output
Temperature change | 15 minutes
  Temperature change
Temperature change | 1 hour
  Temperature change
Temperature change | 2 hours
  Temperature change
Daily fluid balance | 24 hours
  Fluid balance
Daily fluid balance | 48 hours
  Fluid balance

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cronhjort, MD, PhD, Study Director — maria.cronhjort@ki.se
Locations (2):
- Sweden (2):
  - Södersjukhuset, Stockholm
  - Danderyds sjukhus, Stockholm

IPD SHARING:
Plan to Share IPD: No
No data will be shared outside the research group